CLINICAL TRIAL: NCT04028557
Title: Development and Validation of an Integrated Implementation Model for Clinical Decision Support for Heart Failure Prescribing
Brief Title: An Implementation Model for Clinical Decision Support for Heart Failure Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-0020
Record Dates: First submitted 2019-07-08; First posted 2019-07-22 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Decision Support Systems, Clinical; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized CDS (Experimental): The customized CDS will be designed and implemented with comprehensive application of known best practice principles in CDS design. The recommendation will be to initiate an evidence-based beta blocker for heart failure.
  Interventions: Other: Decision Support Systems, Clinical
- Commercial CDS (Active Comparator): The commercial CDS is available to all institutions using the Epic electronic health record vendor, but violates some CDS design best practices, notably not being tailored to the end users of a given health system. The recommendation will be to initiate an evidence-based beta blocker for heart failure.
  Interventions: Other: Decision Support Systems, Clinical

INTERVENTIONS:
Other: Decision Support Systems, Clinical — Active computerized clinical decision support alert within the electronic health record that recommends initiation of an evidence-based beta blocker for heart failure and reduced ejection fraction.
  Other Names: CDS

SUMMARY:
The objective of this proposal is to compare clinical outcomes, implementation metrics (i.e., patient reach and clinician adoption), and clinician preferences of two designs (customized vs. commercial) of a clinical decision support (CDS). Beta blocker prescribing for patients with heart failure will be used as a test case. The best practices in CDS design, including the user-centered design will be incorporated into the customized CDS and compared to a commercially-available CDS in the electronic health record using a cluster randomized trial.

ELIGIBILITY:
Study subjects are providers

Inclusion Criteria:

* Prescribing primary care clinicians at University of Colorado Health (UCHealth) who provide care for patients with heart failure and reduced ejection fraction

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Change in prescription of Beta blocker (BB) | 6 months post CDS implementation
  Number of prescriptions of an evidence based BB during a primary care office visit.

SECONDARY OUTCOMES:
Patient Reach | 6 months post CDS implementation
  The proportion of unique patients with heart failure who were seen by primary care and not taking an evidence based BB who the CDS fired for.
Clinician Adoption | 6 months post CDS implementation
  The proportion of CDS who were not outright dismissed by the clinician.
Factors Influencing Clinician Adoption of the CDS per Qualitative Interviews | 6 months post CDS implementation
  Clinician-reported factors that influence adoption of the CDS.

CONTACTS AND LOCATIONS:
Overall Officials: Katy E Trinkley, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trinkley KE, Kroehl ME, Kahn MG, Allen LA, Bennett TD, Hale G, Haugen H, Heckman S, Kao DP, Kim J, Matlock DM, Malone DC, Page Nd RL, Stine J, Suresh K, Wells L, Lin CT. Applying Clinical Decision Support Design Best Practices With the Practical Robust Implementation and Sustainability Model Versus Reliance on Commercially Available Clinical Decision Support Tools: Randomized Controlled Trial. JMIR Med Inform. 2021 Mar 22;9(3):e24359. doi: 10.2196/24359. PMID 33749610